CLINICAL TRIAL: NCT00295789
Title: A Randomized Phase III Trial of Paclitaxel Plus Cisplatin Versus Paclitaxel Plus Carboplatin in Stage IVb, Persistent, or Recurrent Cervical Cancer (JCOG0505, CC-TPTC-P3)
Brief Title: Trial of TP Versus TC Regimens for Stage IVb, Persistent, or Recurrent Cervical Cancer (JCOG0505, CC-TPTC-P3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0505; C000000335 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Uterine Cervical Neoplasms
Keywords: cervical cancer; palliative chemotherapy; recurrent; persistent; stageⅣb; cisplatin; carboplatin; paclitaxel
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Drug: chemotherapy: Paclitaxel/Cisplatin
  Interventions: Drug: chemotherapy: Paclitaxel/Cisplatin
- 2 (Experimental): Drug: chemotherapy: Paclitaxel/Carboplatin
  Interventions: Drug: chemotherapy: Paclitaxel/Carboplatin

INTERVENTIONS:
Drug: chemotherapy: Paclitaxel/Cisplatin — Drug: chemotherapy: Paclitaxel/Cisplatin
  Arms: 1
Drug: chemotherapy: Paclitaxel/Carboplatin — Drug: chemotherapy: Paclitaxel/Carboplatin
  Arms: 2

SUMMARY:
To evaluate the clinical benefits of Paclitaxel plus Carboplatin compared with Paclitaxel plus Cisplatin in Stage IVb, Persistent, or Recurrent Cervical Cancer

DETAILED DESCRIPTION:
Prognosis of the advanced, recurrent, or persistent cervical cancer, which is not amenable to curative treatment with surgery and/or radiation therapy, still remains poor. Recently, cisplatin plus paclitaxel for palliative chemotherapy were reported to improve the response rate and progression-free interval compared to cisplatin alone and has been shown as a new appropriate regimen. However, more effective and/or less toxic combinations are needed. Carboplatin as a single agent has less response rate but less overall toxicity than cisplatin. Particularly, because less nephrotoxicity does not require hydration and less neurotoxicity enables 3hrs administration of paclitaxel in the combination, out patient therapy becomes possible and patients' quality of life must improve. Therefore, we planned to evaluate the benefits of less toxicity of the chemotherapy containing paclitaxel and carboplatin, which could reduce the hospitalised days, in comparison with the standard chemotherapy containing paclitaxel and cisplatin. This clinical trial is targeted on the patients in Japan with incurable cervical cancer diagnosed by means of image.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven uterine cervical cancer
2. squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the uterine cervix
3. one of the followings, 1)primary stage Ⅳb cervical cancer, 2)the first relapse or persistent cervical cancer after curative first line treatments, 3)the second relapse or persistent cervical cancer after curative second line treatments including radiation, systemic chemotherapy, hormonal therapy, or vaccination therapy for the first relapse
4. Patients may have been previously treated with less than 50 Gy of palliative radiation therapy
5. Patients have received no prior treatment or a certain interval must have elapsed from the last administration of previous treatments including palliative radiation therapy
6. one of the followings, 1)There is at least one metastatic lesion outside the pelvic cavity except paraaortic LN and/or inguinal LN, 2)There is no metastatic lesion outside the pelvic cavity except paraaortic LN and/or inguinal LN and some of the lesions have been irradiated, 3)All lesions are localized inside the pelvic cavity, and some of them have been irradiated
7. no prior surgical therapy for metastatic lesions of the lung or inside the pelvic cavity
8. no bilateral hydronephrosis
9. no prior chemotherapy including more than two platinum-containing regimens
10. no prior chemotherapy including taxane
11. age: 20 to75 years
12. PS: 0-2
13. ANC ≧1,500 /mm3, Plt≧10.0×104/mm3, T-bil≦1.5 mg/dl, GOT（AST）≦100IU/l, sCre ≦1.2 mg/dl, Ccr≧50ml/min in using the Cockcroft-Gault equation, and normal ECG
14. written informed consent

Exclusion Criteria:

1. patients who have some neurologically functional disorder
2. symptomatic CNS metastasis
3. hypersensitive to alcohol
4. active infection
5. HBs antigen positive
6. uncontrollable hypertension
7. history of myocardiac infarction within six months
8. unstable angina
9. uncontrollable diabetes
10. Patients with a concomitant or prior invasive malignancy (except intramucosal malignancy which are curable with local therapy) who have had any evidence of the disease within the last 5 years
11. women during pregnancy or breast-feeding
12. patients with psychiatric illness
13. patients who have been treated with the systemic steroids medication

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2006-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
overall survival | During the study conduct

SECONDARY OUTCOMES:
progression-free survival | During the study conduct
response rate | During the study conduct
adverse events | During the study conduct
severe adverse events | During the study conduct
proportion of periods of non-hospitalization to those of the planned treatment | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiharu Kamura, MD, PhD, Study Chair — Kurume University School of Medicine
Locations (30):
- Japan (30):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Nagoya Medical Center, Nagoya,Naka-ku,Sannomaru,4-1-1, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kyushu University Hospital, Fukuoka,Higashi-ku,Maidashi,3-1-1, Fukuoka
  - National Kyushu Cancer Center, Fukuoka,Minami-ku,Notame,3-1-1, Fukuoka
  - Kurume University School of Medicine, Kurume, Asahi-machi, 67, Fukuoka
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - National Hospital Organization Kure Medical Center Chugoku Cancer Center, Kure,Aoyama-cho,3-1, Hiroshima
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Sapporo Medical University, S-1,W-16,Chuo-ku,Sapporo, Hokkaido
  - Hyogo Medical Center for Adults, Akashi,Kitaouji-cho,13-70, Hyōgo
  - Institute of Clinical Medicine,Tsukuba University Hospital, Tsukuba,Tennodai,1-1-1, Ibaraki
  - Kagoshima City Hospital, Kagoshima,Kajiya-cho,20-17, Kagoshima-ken
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Sinshu University, Matsumoto,Asahi,3-1-1, Nagano
  - Nagaoka Red Cross Hospital, Nagaoka,Terashima-cho,297-1, Niigata
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Osaka City General Hospital, Osaka,Miyakojima-ku,Miyakojimahondori,2-13-22, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - Faculty of Medicine, Saga University, Saga,Nabeshima,5-1-1, Saga-ken
  - Saitama Medical Center, Saitama Medical School, Kawagoe,Komoda,1981, Saitama
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - National Defense Medical College, Tokorozawa,Namiki,3-2, Saitama
  - Juntendo University School of Medicine, Bunkyo-ku,Hongo,3-1-3, Tokyo
  - The University of Tokyo Hospital, Bunkyo-ku,Hongo,7-3-1, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - Jikei University Hospital, Minato-ku,Nishishinbashi,3-25-8, Tokyo
  - Tottori University School of Medicine, Yonago,Nishimachi,36-1, Tottori

REFERENCES:
- [Derived] Kitagawa R, Katsumata N, Shibata T, Kamura T, Kasamatsu T, Nakanishi T, Nishimura S, Ushijima K, Takano M, Satoh T, Yoshikawa H. Paclitaxel Plus Carboplatin Versus Paclitaxel Plus Cisplatin in Metastatic or Recurrent Cervical Cancer: The Open-Label Randomized Phase III Trial JCOG0505. J Clin Oncol. 2015 Jul 1;33(19):2129-35. doi: 10.1200/JCO.2014.58.4391. Epub 2015 Mar 2. PMID 25732161
- See also: Related Info — http://www.jcog.jp/